CLINICAL TRIAL: NCT07396688
Title: Comparative Evaluation of the Effects of Calcium Hydroxide and BIO-C Temp Medicaments on Postoperative Pain in Patients Undergoing Endodontic Treatment: a Clinical Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Assist.Prof.Emine ODABAŞI TEZER, Assistant Professor, Ankara University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 25-AKD-303
Record Dates: First submitted 2026-01-27; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Postoperative Pain; Medicaments Substances in Therapeutic Use; Calcium Hydroxide; Root Canal Retreatment
Keywords: Visual Analog Scale; Postoperative Pain; Bioceramic Intracanal Medicament; Endodontic Retreatment; Calcium Hydroxide
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of two parallel groups according to the intracanal medicament used during the interappointment period. One group receives calcium hydroxide, while the other group receives Bio-C Temp. Each participant is assigned to only one treatment group, and outcomes are evaluated and compared between the two groups over the same follow-up period.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and outcome assessors are blinded to the intracanal medicament used. The intracanal medicaments are applied by a separate investigator who is aware of the treatment assignment but is not involved in outcome assessment or data analysis. Outcome assessments are performed using coded patient records to maintain blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bio-C Temp Group (Experimental): Patients receive Bio-C Temp, a bioceramic-based intracanal medicament, placed in the root canal system during the interappointment period of multi-visit endodontic retreatment.
  Interventions: Drug: bioceramic based intracanal medication
- Calcium Hydroxide Group (Active Comparator): Patients receive calcium hydroxide as an intracanal medicament placed in the root canal system during the interappointment period of multi-visit endodontic retreatment.
  Interventions: Drug: Calcium Hydroxide Intracanal medication

INTERVENTIONS:
Drug: bioceramic based intracanal medication — Bioceramic intracanal medicament (Bio-C Temp®, Angelus):
  A bioceramic-based intracanal medicament used between treatment sessions.
  Arms: Bio-C Temp Group
Drug: Calcium Hydroxide Intracanal medication — Calcium Hydroxide:
  A conventional intracanal medicament used between treatment sessions.
  Arms: Calcium Hydroxide Group

SUMMARY:
This clinical study is designed to evaluate postoperative pain experienced by patients undergoing multi-visit endodontic retreatment and to investigate whether the choice of intracanal medicament influences pain levels between treatment sessions. Postoperative pain is a common concern following root canal procedures and may negatively affect patient comfort, treatment satisfaction, and overall perception of dental care.

Calcium hydroxide has long been used as a conventional intracanal medicament in endodontic therapy due to its antimicrobial properties. In recent years, bioceramic-based materials such as Bio-C Temp have been introduced as alternative intracanal medicaments, with proposed advantages related to biocompatibility and interaction with dental tissues. However, limited clinical evidence is available regarding their effect on postoperative pain when compared with conventional materials.

In this study, patients requiring multi-visit endodontic retreatment will receive either calcium hydroxide or Bio-C Temp as an intracanal medicament between treatment sessions. Pain intensity will be evaluated at specific time points following treatment using standardized pain assessment scales. In addition to pain intensity, the use of analgesic medication will also be recorded.

The primary objective of this study is to compare interappointment postoperative pain levels associated with calcium hydroxide and Bio-C Temp. Secondary objectives include evaluating analgesic consumption. By comparing a conventional intracanal medicament with a newer bioceramic-based alternative, this study aims to contribute to a better understanding of how intracanal medicament selection may influence postoperative pain and patient experience during endodontic retreatment.

The findings of this study may help clinicians make more informed decisions regarding intracanal medicament selection and improve pain management strategies in endodontic practice.

DETAILED DESCRIPTION:
This clinical study is a comparative investigation designed to evaluate interappointment postoperative pain in patients undergoing multi-visit endodontic retreatment. Postoperative pain is a frequent concern in endodontic practice and may affect patient comfort, treatment compliance, and overall satisfaction. The study focuses on whether the choice of intracanal medicament used between treatment sessions influences postoperative pain levels and patient-reported outcomes.

Study Design

The study is conducted as a clinical, comparative study involving patients who require multi-visit endodontic retreatment of single-rooted teeth. Following the initial treatment session, eligible patients are assigned to receive one of two intracanal medicaments during the interappointment period.

Participants

Patients included in the study are systemically healthy individuals classified as ASA Physical Status I, presenting with single-rooted teeth requiring endodontic retreatment and exhibiting normal root anatomy. Patients with conditions or factors that could influence pain perception or treatment outcomes are excluded. All participants provide informed consent prior to enrollment.

Interventions

After completion of the initial endodontic retreatment procedures, intracanal medicaments are placed between treatment sessions. Patients receive either calcium hydroxide, a conventional intracanal medicament, or Bio-C Temp, a newer bioceramic-based intracanal medicament proposed as an alternative to traditional materials. The assigned medicament remains in the root canal system throughout the interappointment period until the subsequent treatment session.

Follow-up and Pain Assessment

Postoperative pain is assessed during the interappointment period using standardized pain assessment tools. Patients are asked to record their pain intensity at predefined time points following the initial treatment session, specifically at 12 hours, 24 hours, 3 days, 5 days, and 7 days. Pain intensity is evaluated using validated pain rating scales, such as the Visual Analog Scale or Numerical Rating Scale.

In addition to pain intensity, patients are monitored for analgesic consumption during the interappointment period. Information regarding the use of pain-relieving medications is recorded at the same follow-up time points.

Outcome Measures

The primary outcome measure of the study is interappointment postoperative pain intensity associated with each intracanal medicament. According to the clinical protocol, a standard-dose analgesic will be prescribed to all participants for postoperative pain control (for example, ibuprofen 400-600 mg to be taken as needed, no more often than every 4-6 hours). Analgesic use will be entirely determined by pain levels, and the number of tablets taken will be documented as a secondary outcome measure.

Study Objective

The primary objective of this study is to compare the effects of calcium hydroxide and Bio-C Temp on interappointment postoperative pain in multi-visit endodontic retreatment. By comparing a conventional intracanal medicament with a newer bioceramic-based alternative, the study aims to provide clinically relevant information that may assist clinicians in selecting intracanal medicaments and improving pain management strategies in endodontic practice.

ELIGIBILITY:
Inclusion Criteria:

* • Patients with single-rooted teeth requiring endodontic retreatment.

  * Individuals in good general health, classified as ASA Physical Status I.
  * Teeth presenting normal anatomical structure and root morphology.

Exclusion Criteria:

* • Patients who have used antibiotics or analgesic medications within the last month.

  * Pregnant individuals and patients with systemic diseases (such as chronic illnesses, diabetes mellitus, hypertension).
  * Teeth with root fractures or perforations.
  * Teeth with complex root canal anatomy, multirooted teeth, or severely curved roots.
  * Patients presenting with high baseline pain levels, particularly those with a history of treatment-resistant pain.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02-10 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Interappointment Pain Intensity | 12 hours, 24 hours, 3 days, 5 days, 7 days
  * What is measured: Postoperative pain intensity will be measured using a patient-reported Visual Analog Scale (VAS).
  * Instrument and range: The VAS is a 10 cm line anchored at 0 cm ("no pain") and 10 cm ("worst possible pain"); participants mark their pain level on this line .
  * Unit and interpretation: Scores range from 0 to 10; higher scores indicate a worse outcome (more pain). The unit of measure is VAS score (0-10).

SECONDARY OUTCOMES:
Analgesic Consumption | Up to 24 hours post-treatment; up to 3 days post-treatment; up to 5 days post-treatment; up to 7 days post-treatment.
  * What is measured: The number of analgesic tablets used by participants for postoperative pain control will be recorded.
  * How measured: At each specified time frame, participants will report the total number of tablets taken since the previous reporting point; values may range from 0 (no analgesics taken) to the maximum number permitted for that interval.
  * Unit and interpretation: The unit of measurement is the number of tablets. Fewer tablets indicate better pain control (less pain).

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University Faculty of Dentistry, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to ethical and confidentiality considerations.

REFERENCES:
- [Background] Wagh KS, Warhadpande MM, Dakshindas DM. Prevalence of endodontic flare-up following intracanal medicament placement in permanent teeth undergoing endodontic treatment - A systematic review. J Conserv Dent. 2022 Jan-Feb;25(1):3-8. doi: 10.4103/jcd.jcd_332_21. Epub 2022 May 2. PMID 35722066
- [Background] Karaoglan F, Kiziltas Gul A, Caliskan MK. Postoperative Pain Following Single-Visit Versus Two-Visit Endodontic Retreatment - A Comparison of Inter-Appointment and Post-Obturation Periods: Randomised Clinical Trial. Aust Endod J. 2025 Dec;51(3):706-714. doi: 10.1111/aej.70004. Epub 2025 Aug 13. PMID 40801476
- [Background] Angin AE, Ozkan HD, Saral IP, Aydin B. The incidence and intensity of postoperative pain and Flare-up following the use of three different intracanal medicaments in teeth with posttreatment apical periodontitis: a randomized clinical trial. Clin Oral Investig. 2024 Jun 8;28(7):362. doi: 10.1007/s00784-024-05760-w. PMID 38849655
- [Background] Omaia M, Negm M, Nashaat Y, Nabil N, Othman A. The effect of triple antibiotic paste as an intracanal medicament with an anti-inflammatory agent on post-operative pain of asymptomatic uniradicular necrotic teeth: a double blind randomized clinical trial. F1000Res. 2025 Dec 16;8:1687. doi: 10.12688/f1000research.19699.3. eCollection 2019. PMID 41552268